CLINICAL TRIAL: NCT00823381
Title: Effect of Resvida(tm) Dietary Supplementation on Muscle Gene Expression: A Comparison With Calorie Restriction Regimen
Brief Title: Effect of Resvida, a Comparison With Calorie Restriction Regimen
Acronym: Resvida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2007-09-25-RESV
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Metabolic Syndrome; Diabetes; Aging
Keywords: obesity; metabolic syndrome; diabetes; aging; calorie restriction; resveratrol; antioxidant
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus | interventions — Resveratrol; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resveratrol (Experimental)
  Interventions: Dietary Supplement: resveratrol
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- Calorie Restriction (Active Comparator)
  Interventions: Behavioral: Calorie Restriction

INTERVENTIONS:
Dietary Supplement: resveratrol — one pill of resveratrol (Resvida™) 75 mg once a day with breakfast
  Other Names: Resvida™
  Arms: Resveratrol
Other: placebo — one placebo pill taken once a day with breakfast
  Arms: Placebo
Behavioral: Calorie Restriction — supervised calorie restriction diet: 30% reduction in caloric intake
  Arms: Calorie Restriction

SUMMARY:
The purpose of this study is to compare the effects of the antioxidant "resveratrol" to a diet intervention (Calorie Restriction) to determine how each of them affects the following: gene expression profile, cholesterol (lipids), how well the hormone insulin works to control your blood sugar, and other blood and tissue markers of metabolic and cardiovascular health.

Resveratrol is found in grape skin, wine, peanuts, and mulberries and is thought to have health benefits such as improving fat metabolism, insulin action, and possibly extending lifespan. Resvida™ is the name for the dietary supplement containing the natural antioxidant "resveratrol". Resvida™ will be supplied by DSM Nutritional Products, Ltd.

Resvida™ is considered a dietary supplement, and therefore it is not an approved drug by the Food and Drug Administration (FDA). It is regulated like a food. The U.S. Food and Drug Administration does not strictly regulate herbs and dietary supplements. The makers of Resvida™ make no claim that this supplement is meant to treat any ailment.

Calorie restriction (CR) is a low calorie diet (about 30% fewer calories than the American Dietetic Association (ADA) recommends). Calorie restriction has also been linked to health benefits (enhanced cardiovascular and metabolic health) and an extended lifespan.

This study is designed to compare the health benefits of both resveratrol and CR and to determine if resveratrol mimics some of the health benefits shown with CR.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females (at least 1 year since last spontaneous menstrual bleeding)
* Caucasian
* Weight (defined as BMI): ≥ 20kg/m2 and < 30 kg/m2.
* Subjects willing and able to give written informed consent and to understand, to participate and to comply with the study requirements with specific agreement to a measurement of global gene expression profiles
* Subjects with the ability to comprehend and complete forms in English
* Subjects who are likely to comply with study procedures
* Subjects who are willing to be assigned to the Resveratrol or CR or Placebo intervention

Exclusion Criteria:

* History of serious or unstable medical or psychiatric disorders (e.g. diabetes, metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic, musculoskeletal, or cancer) that, in the opinion of the investigator, would make the candidate ineligible for the study.
* History of major abdominal, thoracic or non-peripheral vascular surgery within one year prior to the randomization date
* Subjects with any allergic reaction or sensitivity to grape products or any component of the test article
* Subjects who are allergic to lidocaine
* Subjects currently on a low-calorie diet, a weight control or maintenance program, or those who practice a vegetarian or vegan diet
* Subjects who engage in programmed exercise > 2 hours total per week
* Subjects who are smoking or stopped smoking within the past 6 months
* Subjects who have lost or gained >5 kg over the past six months
* Subjects on any other clinical trial or experimental treatment within the past 3 months
* Intake of dietary supplements except vitamins and minerals
* Unwilling to restrict high resveratrol-containing foods
* Current alcohol consumption >20 grams/day
* Current use of the following medications: weight loss medications (prescription or over-the-counter), beta-blockers, steroids, anticoagulants, any other medications that, in the opinion of the investigator, may compromise the validity or safety of the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
global skeletal muscle gene expression profile | three months

SECONDARY OUTCOMES:
insulin sensitivity | three months
intrahepatic triglyceride content, body composition | three months
blood lipid levels, markers of inflammation and plasma hormones | three months
safety and tolerability | three months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States